CLINICAL TRIAL: NCT00397683
Title: Proprietary Information - Exploratory (Non-Confirmatory) Trial
Brief Title: A 52-Week Study to Assess the Effects of MK0822 on Knee Osteoarthritis (MK-0822-011)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-011; 2006_517
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — odanacatib

INTERVENTIONS:
Drug: MK0822

SUMMARY:
The purpose of this study is to test MK0822 on disease activity in patients with osteoarthritis in the knee. Disease modifying activity of MK0822 will be assessed by measurements of knee cartilage using Magnetic Resonance Imaging (MRI) of the knee.

This is an early phase trial and some specific protocol information is proprietary and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic knee osteoarthritis for at least 6 months based on clinical and radiographic criteria
* Patients should be in general good health and must have a certain level of knee pain or be taking pain medicines on most days
* Specific radiographic (X-ray) and MRI features must also be satisfied

Exclusion Criteria:

* Non-osteoarthritic causes of knee pain
* Ineligibility to undergo MRI of the knee due to patient tolerability or safety reasons
* Previous septic arthritis, tibial osteotomy or knee replacement in both knees
* Acute injury of knee ligaments or meniscus in past 2 years
* Knee arthroscopy in past 12 months
* Anticipated arthroscopy or surgery in next 18 months
* Use of intra-articular injections of hyaluronan (e.g. Hyalgan (TM), Synvisc (TM), Orthovisc (TM)) in past 6 months, or injections of glucocorticoids (e.g. Kenalog (TM), Aristospan (TM), Depo-Medrol (TM)) in past 3 months or anticipated knee injections during the study
* Glucosamine or chondroitin sulfate are allowable if they are at a stable dose for past 3 months and will continue at that dose during the study
* Other exclusion criteria apply-Please ask the study doctor for details

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Proprietary Information - Exploratory (Non-Confirmatory) Trial

SECONDARY OUTCOMES:
Proprietary Information - Exploratory (Non-Confirmatory) Trial

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC
Locations (14):
- United States (10):
  - Call for Information, Palm Desert, California
  - Call for Information, Pomona, California
  - Call for Information, Torrance, California
  - Call for Information, Upland, California
  - Call for Information, Coral Gables, Florida
  - Call for Information, Hialeah, Florida
  - Call for Information, South Miami, Florida
  - Call for Information, Rochester, New York
  - Call for Information, Norristown, Pennsylvania
  - Call for Information, Perkasie, Pennsylvania
- Merck Sharp & Dohme (I.A.) Corp., Santiago, Chile
- Frosst Laboratories Inc., Bogota, Cundinamarca, Colombia
- Merck Sharp & Dohme De Mexico, S.A. De C.V., México, D.f., Mexico
- MSD Polska Sp. z o.o. Dzial Medyczny, Warsaw, Poland